CLINICAL TRIAL: NCT03768102
Title: Comparative Study of Verbal Rating Scale and Numerical Rating Scale in Post Anesthesia Care Unit
Brief Title: Comparison of Verbal Rating Scale and Numerical Rating Scale in Post Anesthesia Care Unit
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: SNUMR2-3
Record Dates: First submitted 2018-11-30; First posted 2018-12-07 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Pain Measurement; Acute Pain; Postoperative Pain
MeSH Terms: conditions — Acute Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the postanesthetic care unit(PACU), patients who are recovering from anesthesia are not easy to communicate with. Accordingly, accurate evaluation of acute surgical pain is difficult for PACU patients in spite of severe postoperative pain. Therefore, pain evaluation is clinically important and challenging in PACU. The pain evaluation tool should be simple and easy to understand for accurate assessment. Among the most commonly used pain assessment methods are numerical rating scale(NRS), visual analogue scale(VAS) and verbal rating scale(VRS). These three methods have proved valid for clinical situations in many studies. VRS appears to be easier to understand than the other two methods for patients in PACU. The purpose of this study is to compare NRS and VRS in PACU patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent general anesthesia
* The American Society of Anesthesiologists(ASA) physical status classification system : class 1, 2, 3

Exclusion Criteria:

* The American Society of Anesthesiologists(ASA) physical status classification system : class 4, 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An adult patient who has been transferred to the recovery room after receiving general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Pain measurement by the numerical rating scale | 5 minutes after transferred into the postanesthesia care unit
  Patients verbally requested to rate their pain : "Rate your pain from 0 (no pain) to 10 (unbearable pain)".
  0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
Pain measurement by the numerical rating scale | 20 minutes after transferred into the postanesthesia care unit
  Patients verbally requested to rate their pain : "Rate your pain from 0 (no pain) to 10 (unbearable pain)" 0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
Pain measurement by the numerical rating scale | 40 minutes after transferred into the postanesthesia care unit
  Patients verbally requested to rate their pain : "Rate your pain from 0 (no pain) to 10 (unbearable pain)" 0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
Pain measurement by the verbal rating scale | 5 minutes after transferred into the postanesthesia care unit
  Patients verbally requested to answer which of the four categories you belong to : no pain, mild pain, moderate pain, severe pain
Pain measurement by the verbal rating scale | 20 minutes after transferred into the postanesthesia care unit
  Patients verbally requested to answer which of the four categories you belong to : no pain, mild pain, moderate pain, severe pain
Pain measurement by the verbal rating scale | 40 minutes after transferred into the postanesthesia care unit
  Patients verbally requested to answer which of the four categories you belong to : no pain, mild pain, moderate pain, severe pain
nonresponse rate of the numerical rating scale | 1 year
  the rate of assessment failures among the total number of assessment
nonresponse rate of the verbal rating scale | 1 year
  the rate of assessment failures among the total number of assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Jin-Tae Kim, Seoul, Select, South Korea

IPD SHARING:
Plan to Share IPD: No